CLINICAL TRIAL: NCT05379413
Title: Comprehensive Observational & Longitudinal Study on the Outbreak of Stroke Related Spasticity Focusing on the Early Onset Management With BoNT: The COLOSSEO-BoNT Study
Brief Title: Observational Longitudinal Study on the Outbreak and Management of Stroke Related Spasticity
Acronym: COLOSSEO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Massimo Marano, Principal Investigator, Campus Bio-Medico University
Other Study IDs: COLOSSEO-BoNT
Record Dates: First submitted 2022-05-10; First posted 2022-05-18 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Spasticity as Sequela of Stroke
Keywords: Botulinum neurotoxin type A (BoNT-A); Stroke; Rehabilitation; Post-Stroke Spasticity (PSS)
MeSH Terms: conditions — Stroke | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Early BoNT treatment: Patients with PSS treated with BoNT within the first Quartile of injection timing distribution
  Interventions: Drug: Botulinum toxin type A
- Late BoNT treatment: Patients with PSS treated with BoNT within the third Quartile of injection timing distribution
  Interventions: Drug: Botulinum toxin type A
- Not treated with BoNT: Natural controls with PSS not treated with BoNT

INTERVENTIONS:
Drug: Botulinum toxin type A — Botulinum neurotoxin (BoNT) Type A injection with either OnaBoNT-A, AboBoNT-A, IncoBoNT-A
  Groups: Early BoNT treatment; Late BoNT treatment

SUMMARY:
Stroke is one of the leading cause of death and disability worldwide. Post-stroke spasticity (PSS) is outbreak after a stroke and is featured by disabling muscle stiffness. PSS could manifest in up tp 50% cases within 6 months after a stroke, especially in the upper limb. Despite it is an acknowledged condition it is insufficiently recognized and treated in clinical practice.

Focal and regional spasticity could improve with rehabilitation and in selected cases with botulinum neurotoxin (BoNT) type A injections. The latter causes muscle relaxation and fosters neuroplasticity, which is able in turn of ameliorating several patient functional aspects. Recent literature demonstrated that PSS patients treated with early BoNT (within 3 month since PSS outbreak) could improve in their clinical status better than patients with a later treatment.

An earlier recognition of PSS predictors could improve patient management. Hence, the investigators are going to perform a multicentric prospective observational real life study with BoNT, based on the best clinical practice and aimed at the early recognition and management of PSS through the identification of 1) early clinical predictors of spasticity (collected within 10 days since stroke), 2) BoNT clinical outcome relative to the timing of the treatment

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke with onset not far than 10 days before the enrollment
* BoNT naive
* Ability to sign the informed consent

Exclusion Criteria:

* Hypersensitivity to BoNT or BoNT related substances
* Participant of Post-stroke spasticity RCT
* Persistent and severe altered mental status or concurrent severe medical condition able to hasten the rehabilitation path.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients suffering for ischemic stroke with upper limb involvement treated at the Lazio region (Italy) stroke units.
Sampling Method: Non-Probability Sample
Enrollment: 960 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Upper limb post stroke-spasticity development | 0-24 months
  Detection of a Modified Ashworth Scale (MAS) >/= 1 at the upper limb (MAS is a 0 to 5 score, with score 5 as the worst rigidity possible)

SECONDARY OUTCOMES:
Post-Stroke Spasticity in early vs late treatment | 3-24 months
  Comparison of the Modified Ashworth Scale (MAS) at the elbow and wrist (MAS is a 0 to 5 score, with score 5 as the worst rigidity possible) in early versus late treatment

OTHER OUTCOMES:
Upper limb functionality | 3-24 months
  Comparison of functional items of upper limb functionality (arm activity measure scale, i.e. ARM-A a 0-84 scale - a higher score means a worse upper limb function) of early versus late treatments
Quality of Life measurement | 3-24 months
  Comparison of Quality of Life (EuroQoL-5D or EQ-5D scale , 5 to 25 scale where 25 is the worst quality of life possible) of patients with early versus late treatments
Pain measurement | 3-24 months
  Comparison of pain (Visual Analogue scale or VAS in units on a 0-10 grading system, where 10 is the worst pain possible) of patients with early versus late treatments
Spasticity in Botulinum Toxin (BoNT) treated versus untreated patients | 3-24 months
  Comparison of modified ashworth scale (MAS) in BoNT treated versus untreated subjects (MAS is a 0 to 5 score, where 5 is the worst rigidity possible). Herein an aggregated wrist and elbow score (on a 0 - 10 scale with 10 being the worst spasticity) will be used.
Functionality in Botulinum Toxin treated versus untreated patients | 3-24 months
  Comparison of functionality (arm activity measure, i.e. ARM-A total score, a 0 to 84 scoring system - higher score means a worse upper limb function) in BoNT treated versus untreated subjects
Quality of life in Botulinum Toxin treated versus untreated patients | 3-24 months
  Comparison of Quality of life (EuroQoL-5D or EQ-5D scale is a 5 to 25 scale where 25 is the lower quality of life possible) in BoNT treated versus untreated patients
Pain in Botulinum Toxin treated versus untreated patients | 3-24 months
  Comparison of pain (visual analogue scale, VAS, 0-10 scale where 10 is the worst pain possible) in BoNT treated versus untreated patients

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - ASL RM 1 San Filippo Neri Hospital, Rome, Lazio
  - Sapienza University of Rome - Stroke Unit, Rome, Lazio
  - Sapienza University of Rome, Rome, Lazio
  - Fondazione Policlinico Universitario Campus Bio-Medico, Rome, Lazio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeng H, Chen J, Guo Y, Tan S. Prevalence and Risk Factors for Spasticity After Stroke: A Systematic Review and Meta-Analysis. Front Neurol. 2021 Jan 20;11:616097. doi: 10.3389/fneur.2020.616097. eCollection 2020. PMID 33551975
- [Background] Wissel J, Fheodoroff K, Hoonhorst M, Mungersdorf M, Gallien P, Meier N, Hamacher J, Hefter H, Maisonobe P, Koch M. Effectiveness of AbobotulinumtoxinA in Post-stroke Upper Limb Spasticity in Relation to Timing of Treatment. Front Neurol. 2020 Feb 28;11:104. doi: 10.3389/fneur.2020.00104. eCollection 2020. PMID 32184753
- [Background] Picelli A, Santamato A, Cosma M, Baricich A, Chisari C, Millevolte M, Prete CD, Mazzu I, Girardi P, Smania N. Early Botulinum Toxin Type A Injection for Post-Stroke Spasticity: A Longitudinal Cohort Study. Toxins (Basel). 2021 May 24;13(6):374. doi: 10.3390/toxins13060374. PMID 34073918
- [Background] Opheim A, Danielsson A, Alt Murphy M, Persson HC, Sunnerhagen KS. Early prediction of long-term upper limb spasticity after stroke: part of the SALGOT study. Neurology. 2015 Sep 8;85(10):873-80. doi: 10.1212/WNL.0000000000001908. Epub 2015 Aug 14. PMID 26276377
- [Derived] Marano M, Suppa A, Palmieri MG, Cecconi E, Frisullo G, Bovenzi R, Riso V, Anzini A, Brienza M, Anticoli S, Crupi D, Giovannelli M, Massimiani A, Rinalduzzi S, Morena E, Massara MC, Cupini L, Bressi F, Pilato F, Maggi L, Sauchelli D, Iezzi E, Centonze D, Aprile I, Di Lazzaro V, Toni D, Altavista MC; COLOSSEO study group. Comprehensive Observational and Longitudinal study on the Outbreak of Stroke-related Spasticity focusing on the Early Onset management with Botulinum NeuroToxin (COLOSSEO-BoNT): protocol for a real-world prospective observational study on upper limb spasticity. BMJ Open. 2024 Jul 1;14(6):e085484. doi: 10.1136/bmjopen-2024-085484. PMID 38950995